CLINICAL TRIAL: NCT02556619
Title: Early Symptom Control and Palliative Care Referral for Advanced Hepatocellular Carcinoma; a Randomized Control Trial
Brief Title: Randomized Control Trial (RCT) of Early Palliative Care for HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Curtis Jackson Wray, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-15-0559
Record Dates: First submitted 2015-09-10; First posted 2015-09-22 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Liver Cancer; Randomized Control Trial; Palliative Care; Liver Cell Carcinoma; Palliative Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapy (No Intervention): Patients will undergo standard medical care for Hepatocellular Carcinoma diagnosis.Patients however will not be denied early palliative care if requested.
- Early Palliative Care/Symptom Control (Experimental): Patients will undergo palliative care services at time of Hepatocellular Carcinoma diagnosis.
  Palliative care and symptom control services are adapted from the National Consensus Project for Quality Palliative Care.
  Early referral, patients meeting inclusion criteria will be enrolled and referred to palliative care within 3 weeks of the index consultation with Medical-Oncology, Surgical-Oncology or Gastroenterology.
  Intervention will be:
  1. Establish palliative care goals
  2. Symptom Assessment and Control
  3. End-of-Life Care
  Interventions: Behavioral: Early Palliative Care/Symptom Control

INTERVENTIONS:
Behavioral: Early Palliative Care/Symptom Control — 1. Establish palliative care goals
     1. Determination of Medical Power of Attorney
     2. Discuss/plan code status/advance directives
     3. Document palliative care goals
  2. Symptom Assessment and Control
     1. Pain-treatment with opioid and non-opioid medications
     2. Itching-H2 blockers, steroids
     3. Nutrition-appetite stimulated with Megace, review low sodium diet
     4. Ascites/edema- optimize ascites management with Lasix or Aldactone. In refractory cases intermittent paracentesis can be performed
     5. Nausea- treated with anti-emetics
     6. Jaundice and Body Image- counselling regarding symptoms
  3. End-of-Life Care
     1. Discuss religious preferences
     2. Assess for distress- ensure interaction with Cancer Resource Center
     3. Hospice- charity Hospice options for select patients.
  Arms: Early Palliative Care/Symptom Control

SUMMARY:
The purpose of this research study is to evaluate the effect of early palliative care consultation on quality of life, use of hospital resources, end-of-life care and survival among Hepatocellular Carcinoma (HCC) patients with advanced End Stage Live Disease not eligible for potentially curative or local area therapy. Half of patients will receive early palliative care at diagnosis of HCC and other half will receive palliative care when all standard therapy treatments have been exhausted.

DETAILED DESCRIPTION:
Intro:

Hypothesis Methods Analysis Anticipated Results

Palliative care will focus on providing relief from the symptoms and stress associated from cancer. This helps improve quality of life for cancer patients and their family. This care is usually offered to patients when all standard therapy treatments have been exhausted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed HCC by biopsy or liver protocol CT scan or MRI characteristics
* Permanent street address with Harris County, Texas and consent to study participation
* English or Spanish speaking with ability to respond to the QoL questionnaires
* Child-Pugh C, not eligible for liver transplantation (TXP), surgical resection, ablation, locoregional or systemic therapy
* Child-Pugh C, eligible for systemic chemotherapy (Sorafenib), not eligible for TXP, surgical resection, ablation or locoregional therapy
* Child-Pugh A or B, not eligible for surgical resection or ablation (>3 lesions or 2 lesions with one being >5cm)
* Child-Pugh A, not eligible for TXP, surgical resection, ablation or locoregional therapy

Exclusion Criteria:

* Primary modality of treatment is potentially curative TXP, surgical resection or ablation as deemed by GI MDC
* Child-Pugh A or B (up to 2 lesions < 5cm in size)
* Medical (e.g. severe encephalopathy), psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any medical condition (acute myocardial infarction or stroke) that could jeopardize the safety of the patient and his/her compliance in the study
* Vulnerable population (inmates in jail or prison)
* Non-English or Non-Spanish Speaking patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life (HRQoL) | 6 months
  The primary outcome is the change in the patient's primary need based upon HRQoL survey. These scores range from 0-100 for the role functioning scale, physical function scale and the other QLQ-C30 scales and HCC18 symptom complexes.

SECONDARY OUTCOMES:
Survival | 2 Years after diagnosis
  Overall Survival. The investigators will assess if the intervention improves overall survival. The unit of measure will be months
Resource Utilization | 2 Years after diagnosis
  The investigators will determine if the intervention decreases resource utilization (ICU days and length of stay). The unit of measure will be days.
Cost Utilization | 2 Years after diagnosis
  The investigators will determine if the intervention decreases cost between groups. To do this, the investigators will track cost per group from time of study enrollment to either death, withdrawal or study completion. Cost will be estimated in US dollars.

CONTACTS AND LOCATIONS:
Overall Officials: Curtis J Wray, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Lyndon Baines Johnson (LBJ) General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No